CLINICAL TRIAL: NCT07149792
Title: A Multi-center RCT Clinical Trial on Personalized Precision Medicine for Patients With Psoriasis and Psoriatic Arthritis and Investigation on Cardiovascular Biomarkers
Acronym: SMILE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Chung Shan Medical University (Other); Far Eastern Memorial Hospital (Other); China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Taichung VGH Derm Yen; TCVGH-1445602C (Other Grant/Funding Number: TAICHUNG VETERANS GENERAL HOSPITAL)
Record Dates: First submitted 2025-08-17; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis; Psoriasis Arthritis; Biologics
Keywords: Prescreen, Biologics, Psoriasis, Strategic selection, Psoriatic arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: The psoriasis patients are arranged randomly by two groups:
  1. Strategic groups: This group patients prescreen to various biologics on their immune cells and choose the most proper biologics according to a set of biomarkers for individual psoriasis patient before starting the treatment.
  2. Standard groups: This group patients receive biologics treatment according to present guideline without individual immune cells screen.
  The patients are enrolled need washout bioloigics1 month but dMARD is exceptional. We will collect the clinical data including PASI, BSA, Pruritus score, Swelling joint counts, Tender joint counts, DAPSA score, DLQI score in the follwing timetable to 3 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prescreen Based bDMARD Stategic Treatment Group (Experimental): Strategic groups: This group patients prescreen to various biologics (such as Adalimumab (Humira), Etanercept (Enbrel), Certolizumab pegol (Cimzia) Golimumab (Simponi), Ustekinumab (Stelara),Secukinumab (Cosentyx) Ixekizumab (Taltz),Bimekizumab (Bimzelx), Brodalumab (Lumicef)) on their immune cells and choose the most proper biologics according to a set of biomarkers for individual psoriasis patient before starting the treatment
  Interventions: Diagnostic Test: Prescreen platform; Biological: biologics treatment
- Standard bDMARD Treatment Group (Active Comparator): This group patients receive biologics treatment (such as Adalimumab (Humira), Etanercept (Enbrel), Certolizumab pegol (Cimzia) Golimumab (Simponi), Ustekinumab (Stelara),Secukinumab (Cosentyx) Ixekizumab (Taltz),Bimekizumab (Bimzelx), Brodalumab (Lumicef)) according to present guideline without individuals immune cells screen.
  Interventions: Biological: biologics treatment

INTERVENTIONS:
Diagnostic Test: Prescreen platform — Different biomarkers on PsO, PsA and paradoxical PsA
  Arms: Prescreen Based bDMARD Stategic Treatment Group
Biological: biologics treatment — All psoriasis patients are receiving biologics treatment

SUMMARY:
The inclusion criteria for this study were patients aged 18 to 75 years with a confirmed diagnosis of psoriasis by a dermatologist or psoriatic arthritis by a rheumatologist. Patients with active infections or suspected malignancies were excluded.

A total of 40 patients with psoriasis, with or without psoriatic arthritis, were enrolled from multiple centers in Taiwan. All participants were recruited from the outpatient clinics of either the Department of Allergy, Immunology, and Rheumatology or the Department of Dermatology in tertiary hospitals across Taiwan.

Participants were randomly assigned to one of two groups:

Prescreen Strategy-Based Biologics Selection Group

Standard-Based Biologics Selection Group

Patients will be followed up at weeks 4, 8, 12, 24, 32, 40, 48, 56, 64, and 72. Follow-up may be extended up to 3 years if necessary.

Clinical assessments will include:

Primary endpoints: PASI (Psoriasis Area and Severity Index), painful joint count, swollen joint count, and DAPSA (Disease Activity in Psoriatic Arthritis) score.

Secondary endpoints: DLQI (Dermatology Life Quality Index), BSA (Body Surface Area), pruritus score, and internal carotid artery thickness measured at 6 months, 1 year, and 2 years.

DETAILED DESCRIPTION:
To prepare the PBMC (peripheral blood mononuclear cell) culture, 16 mL of peripheral blood is collected from each patient using sodium citrate tubes (Vacutainer CPT, BD Biosciences, Franklin Lakes, NJ, USA). PBMCs are isolated by centrifugation at 1800 × g for 20 minutes at room temperature with the brake turned off, resulting in the separation of plasma, PBMCs, gel plugs, and red blood cell (RBC) layers.

The isolated PBMCs are washed with phosphate-buffered saline (PBS) and then cultured in RPMI-1640 medium supplemented with 10% fetal bovine serum (FBS) and 1% penicillin/streptomycin at 37 °C in a 5% CO₂ incubator.

A total of 6 × 10⁵ cells/mL are seeded into 12-well plates and treated for 24 hours under the following conditions:

Control

Streptococcus pyogenes only

S. pyogenes + adalimumab (4 μg/mL)

S. pyogenes + golimumab (0.5 μg/mL)

S. pyogenes + certolizumab (20 μg/mL)

S. pyogenes + ustekinumab (0.25 μg/mL)

S. pyogenes + ixekizumab (3.5 μg/mL)

S. pyogenes + secukinumab (16.7 μg/mL or 34 μg/mL)

S. pyogenes + guselkumab (1.2 μg/mL)

S. pyogenes + risankizumab (2 μg/mL)

Culture supernatants are collected for subsequent cytokine measurement. The concentrations of biological agents used correspond to the trough serum concentrations at steady state as indicated in the pharmacokinetic sections of reference data. The two concentrations of secukinumab (16.7 μg/mL and 34 μg/mL) reflect the two common clinical doses of 150 mg and 300 mg per month, respectively.

Cytokine Analysis

Cytokine levels are measured in the collected supernatants using a protein multiplex immunoassay system (Bio-Plex Cytokine Array System, Bio-Rad Laboratories, Hercules, CA, USA). The following cytokines and chemokines are analyzed:

IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12, IL-13, IL-17A, IFN-γ, TNF-α, monocyte chemoattractant protein-1 (MCP-1), macrophage inflammatory proteins (MIP-1α and MIP-1β), platelet-derived growth factor-BB (PDGF-BB), and chemokine (CC motif) ligand 5 (RANTES).

Screening Method for Biologic Agents

RANTES Exclusion First, biologics that induce a RANTES level ≥1.5 times higher than that of S. pyogenes-only treatment are excluded.

Scoring System for Biologic Selection in Psoriasis

Remaining biologics are categorized into three grades based on biomarker levels:

IFN-γ

IL-17A

IFN-γ/IL-4

IFN-γ/IL-13

IL-17A/IL-4

IL-17A/IL-13

Grade 1 (Most appropriate): Lowest biomarker values

Grade 2 (Possibly appropriate): Intermediate values

Grade 3 (Not recommended): Highest values

Each grade is subdivided into a, b, and c groups:

Lower values within a grade are ranked as a, followed by b, then c

Scoring is as follows:

1. a = +3, 1b = +2, 1c = +1.5
2. a = +1, 2b = +0.5, 2c = 0
3. a = -0.5, 3b = -1, 3c = -1.5

The total score for each biologic is the sum of individual biomarker scores. Based on total scores:

High score = Most appropriate

Medium score = Possibly appropriate

Low score = Not recommended

Scoring for Psoriatic Arthritis (PsA)

For PsA, biologics are selected based on the lowest RANTES, MCP-1 and IFN-γ levels:

Grade 1 (Most appropriate): Lowest biomarker values Grade 2 (Possibly appropriate): Intermediate values Grade 3 (Not recommended): Highest values RANTES: 2+, 1+, 0 MCP-1: 1+, 0.5+, 0 IFN-γ: 1+, 0.5+, 0 The final score is the sum of RANTES MCP-1 and IFN-γ scores. Biologics with the lowest total scores are preferred.

Patient Assignment in Strategic Group

Biologics from the "most appropriate" group are selected for each patient in the strategic group. The following clinical indicators are monitored over time:

Absolute PASI

Tender joint count

Swollen joint count

DAPSA score

DLQI

Internal carotid artery intima thickness

Follow-up Timeline

Clinical assessments: Weeks 0, 2, 4, 12, 24, and 48

Intima thickness: Weeks 0 and 48

Outcome Comparison Outcomes between the strategic selection group and standard care group are compared at Weeks 24 and 48, with extended follow-up up to 5 years. Primary outcomes include PASI and DLQI scores.

Statistical Analysis

All statistical analyses are conducted using SPSS version 22 (IBM, Armonk, NY, USA). Demographic and clinical characteristics, as well as outcome measures (PASI, joint counts, DAPSA, DLQI, and carotid intima thickness), are analyzed using the Mann-Whitney U test and Spearman's rho correlation.

Data are presented as mean ± standard deviation. Two-sided p values < 0.05 are considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Psoriasis patients
* Psoriatic arthritis patients
* Agree to provide a blood sample

Exclusion Criteria:

* A current history of cancer,
* Recent hospitalization for infection or current antibiotic treatment
* HIV infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
PASI (Psoriasis Area and Severity Index) | From enrollment to the end of treatment at 48 weeks
  The skin condition of psoriasis patients is assessed using the PASI (Psoriasis Area and Severity Index), which ranges from 0 to 72, with higher scores indicating more severe disease
DAPSA Score - Disease Activity in Psoriatic Arthritis | From enrollment to the end of treatment at 48 weeks
  DAPSA Formula (Total Score):
  DAPSA = TJC (68)
  + SJC (66)
  + Patient Global Assessment (0-10)
  + Patient Pain Assessment (0-10)
  + CRP (mg/dL) DAPSA=TJC (68)+SJC (66)+Patient Global Assessment (0-10)+Patient Pain Assessment (0-10)+CRP (mg/dL)
  Where:
  TJC = Tender Joint Count (out of 68 joints)
  SJC = Swollen Joint Count (out of 66 joints)
  Patient Global Assessment (PtGA) = Patient's rating of overall disease activity (0-10 scale)
  Pain VAS = Patient's self-reported pain (0-10 scale)
  CRP = C-reactive protein level (mg/dL)
  Interpreting DAPSA Scores:
  DAPSA Score and Disease Activity Level
  ≤4 Remission, >4-14 Low disease activity, >14-28 Moderate disease activity, >28 High disease activity

SECONDARY OUTCOMES:
BSA (body surface area) | From enrollment to the end of treatment at 48 weeks
  The severity of psoriatic disease can be assessed using the Body Surface Area (BSA) score, which ranges from 0 to 100%. A higher BSA score indicates more extensive and severe skin involvement
Pruritus score | From enrollment to the end of treatment at 48 weeks
  The severity of psoriatic disease can be assessed using the pruritus score, which ranges from 0 to 10. A higher pruritus score indicates more severe skin involvement
Swelling joint counts | From enrollment to the end of treatment at 48 weeks
  0 swollen joints = No active synovitis (remission or well-controlled disease)
  Higher counts = More active joint inflammation and more severe disease
Tender joint counts | From enrollment to the end of treatment at 48 weeks
  0 tender joints = No current joint pain (remission or well-controlled disease) Higher TJC = Greater disease burden or active joint inflammation
Dermatology Life Quality Index (DLQI) | From enrollment to the end of treatment at 48 weeks
  The DLQI (Dermatology Life Quality Index) score ranges from 0 to 30, with higher scores indicating a greater impact of the disease on the patient's quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taichung Veterans Hospital, Taichung, Taiwan
  - Taichung Vertenans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication